CLINICAL TRIAL: NCT04649203
Title: Multicenter, Double-blind, Placebo-controlled Randomized Clinical Trial of Efficacy and Safety of the Drug Cytoflavin®, Administered Intravenously Followed by Oral Intake, in Patients With Diabetic Polyneuropathy
Brief Title: Cytoflavin in the Treatment of Patients With Diabetic Polyneuropathy
Acronym: CYLINDER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTF-III-DM-2019
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetes Mellitus; Peripheral Nervous System Diseases; Antioxidants; Succinic acid
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Peripheral Nervous System Diseases | interventions — cytoflavin; Inosine; Niacinamide; Riboflavin; Succinic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Cytoflavin (Inosine + Nicotinamide + Riboflavin + Succinic Acid), 20 ml (two ampoules of 10 ml each) once a day intravenously in a dilution of 200 ml of 0.9% sodium chloride solution at a rate 3-4 ml/min, for 10 days + Cytoflavin ((Inosine + Nicotinamide + Riboflavin + Succinic Acid), 2 tablets 2 times a day, for 75 days
  Interventions: Drug: Cytoflavin (Inosine + Nicotinamide + Riboflavin + Succinic Acid)
- Group 2 (Placebo Comparator): Placebo, 20 ml (two ampoules of 10 ml each) once a day intravenously in a dilution of 200 ml of 0.9% sodium chloride solution at a rate 3-4 ml / min, for 10 days + Placebo, 2 tablets 2 times a day, for 75 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cytoflavin (Inosine + Nicotinamide + Riboflavin + Succinic Acid) — The study drug will be administered in two phases: intravenous infusion of study drug for 10 days followed by oral administration of study drug for 75 days. Thus, the total duration of the study therapy is 12 weeks.
  Arms: Group 1
Drug: Placebo — The placebo comparator will be administered in two phases: intravenous infusion of placebo solution for 10 days followed by oral administration of placebo pills for 75 days. Thus, the total duration of the study therapy is 12 weeks.
  Arms: Group 2

SUMMARY:
One of the most common complications of diabetes mellitus is diabetic polyneuropathy, which leads to disability and reduces quality of life. The toxic effects of high glucose concentrations contribute to the formation of ketoaldehyde free radicals, which, at an increased rate of their formation, leads to the development of oxidative stress in the nervous tissue. The planned study of the use of Cytoflavin® in diabetic polyneuropathy is substantiated by its antioxidant effect, which, by analogy with alpha-lipoic acid preparations, suggests its efficacy in the combined treatment of such patients. This clinical study is being conducted to assess the efficacy and safety of Cytoflavin® versus Placebo in diabetic polyneuropathy patients with type 2 diabetes. Study patients will receive study medication, 10 IV infusions followed by 75 days of oral intake. Clinical efficacy will be assessed by alleviation of symptoms (burning, numbness, pain and pricking), using the total symptoms score(TSS), after the completion of the treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Men and women aged 45 to 74 (inclusive);
* Confirmed diagnosis of type 2 diabetes lasting for 1 year or more;
* Permanent scheme of therapy (without changing doses and drugs) by oral hypoglycemic drugs and / or insulin, long-term or ultra-long (adjustment of insulin dose is possible within 10% from baseline dose) and / or agonists of glucagon-like peptide-1 receptors (GLP-1) for at least 12 weeks before screening;
* HbA1c from 7.0 and not higher than 10.0%;
* BMI 22-40 kg / m2;
* Symptomatic distal sensorimotor diabetic polyneuropathy;
* Baseline TSS (Total Syptom Score) ˃5 points;
* Score ≥2 by at least one of the TSS symptoms;
* The severity of pain by the corresponding TSS subscale ≤ 2;
* NISLL (Neuropathy Impairment Score Low Limbs) ≥ 2 points;
* Patient consent to use adequate contraceptive methods for the entire study;
* Consent to maintain a stable diet, exercise, therapy and diabetes control throughout the study;
* Ability to comply with all protocol requirements.

Exclusion Criteria:

* Pregnant or lactating women, or women planning a pregnancy during a clinical trial;
* Type 1 diabetes and other specific types of diabetes;
* Acute metabolic complications of diabetes such as ketoacidosis or hyperosmolar state within 6 months prior to screening;
* Therapy with short and ultra-short insulin within 3 months before screening;
* Fasting plasma glucose at screening> 15 mmol / l;
* The presence of severe complications of diabetes;
* Epilepsy, epileptiform seizures, head trauma with loss of consciousness, tumor, inflammatory and demyelinating diseases of the central nervous system;
* Diseases requiring prior or current treatment by systemic corticosteroid drugs, cytostatics or penicillamine;malignant neoplasms within the last 5 years (excluding basal cell carcinoma);
* Cardiovascular diseases in the stage of decompensation at present or within 3 months before screening;
* Uncontrolled arterial hypertension with systolic arterial pressure> 180 mm Hg and diastolic blood pressure> 110 mm Hg at screening;
* Nephrotic syndrome, severe chronic renal failure or significant kidney disease with a level of glomerular filtration rate (GFR) <30 ml / min;
* Active viral (hepatitis B and C) or cirrhotic liver disease; increased aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT) 3 times from upper normal limit; increased total bilirubin 2 times from upper normal limit;
* HIV; a severe infectious disease within 30 days before screening;
* Anemia (hemoglobin ≤ 105 g / l in women or ≤ 115 g / l in men); acute blood loss or donation of at least one unit of blood (500 ml) or blood transfusion within the previous 12 weeks;
* Drug or alcohol abuse;
* Intake of Cytoflavin® for 3 months before screening;
* Known allergies, hypersensitivity or contraindications to the drug Cytoflavin® or its components;
* Intake of alpha-lipoic acid, thiamine derivatives, pyridoxine, cyanocobalamin (excluding multivitamins), antidepressants and derivatives of gabapentin within 3 months before screening;
* Use of other investigational drugs within 3 months prior to screening;
* Inability to read or write; unwillingness to understand and follow protocol procedures; non-compliance with the protocol requirements.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
TSS (Total Symptom Score) | 12 weeks
  Change in total TSS score at Week 12 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Igor A Strokov, Prof., Study Chair — "First Moscow State Medical University n.a. I.M.Sechenov of the Ministry of Health of Russia
Locations (16):
- Russia (16):
  - City Clinical Hospital n.a. V.P.Demikhov, Moscow
  - City Clinical Hospital n.a.M.E.Zhadkevitch, Moscow
  - City Clinical Hospital #13 Avtozavodsky district, Nizhny Novgorod
  - Research Center for Eco-safety, Ltd., Saint Petersburg
  - "Astarta" Ltd., Saint Petersburg
  - "Consultative and diagnostic center with a polyclinic" of the Administrative Department of the President of the Russian Federation, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - City General Hospital №2, Saint Petersburg
  - City Outpatient Clinic #117, Saint Petersburg
  - City Outpatient Clinic #51, Saint Petersburg
  - I. P. Pavlov 1st St. Petersburg State Medical University, Saint Petersburg
  - MEDICA Ltd., Saint Petersburg
  - North-West State Medical University named after I.I. Mechnikov, Saint Petersburg
  - "Diabetes" medical center, Samara
  - Saratov State Medical University n.a. V.I.Razumovsky, Saratov
  - GBUZ YAO "Regional Clinical Hospital", Yaroslavl

REFERENCES:
- [Result] Kharitonova T, Shvarts YG, Verbovoy AF, Orlova NS, Puzyreva VP, Strokov IA. Efficacy and safety of the combined metabolic medication, containing inosine, nicotinamide, riboflavin and succinic acid, for the treatment of diabetic neuropathy: a multicenter randomized, double-blind, placebo-controlled parallel group clinical trial (CYLINDER). BMJ Open Diabetes Res Care. 2022 Jun;10(3):e002785. doi: 10.1136/bmjdrc-2022-002785. PMID 35680173